CLINICAL TRIAL: NCT05478109
Title: the Material Balance and Biotransformation Study of [14C] XZP-3287 in Healthy Chinese Male Subjects
Brief Title: A Clinical Trial of XZP-3287 for Material Balance
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xuanzhu Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: XZP-3287-1004
Record Dates: First submitted 2022-07-18; First posted 2022-07-28 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Healthy Male Subjects

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C]XZP-3287 (Experimental): Eligible healthy male subjects received a single oral 360 mg (radioactivity of 50µCi) dose of [14C]XZP-3287
  Interventions: Drug: [14C]XZP-3287

INTERVENTIONS:
Drug: [14C]XZP-3287 — 360 mg suspension containing 50µCi of [14C] XZP-3287

SUMMARY:
A single-centre, open-label, mass balance and biotransformation study in healthy male subjects utilising a single oral dose of [14C] XZP-3287

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult males aged 18 to 45 years (inclusive).
2. Body weight ≥ 50 kg for males; body mass index (BMI) in the range 19-26 kg/m2 (inclusive).
3. No mental disorders, cardiovascular system, nervous system, respiratory system, digestive system, urinary system, endocrine system and metabolic abnormalities.
4. No clinically significant vital signs, physical examination, laboratory tests, ECG findings.
5. No plans to have children within the last 12 months, and willing to use effective contraception within 12 months after the end of dosing.
6. Subjects are able to communicate well with the investigators, and be able to complete the trial according to the process, and sign an Informed Consent Form.

Exclusion Criteria:

1. Subjects with a history of drug allergy, or atopic allergic disease (Asthma, urticaria, eczema dermatitis), or a known history of allergy to the test drug or its adjuvant components.
2. History of clinically significant ECG abnormalities or family history of long QT syndrome.
3. History of any significantly diseases affect drug absorption, distribution, metabolism, and excretion.
4. Positive test for hepatitis B (surface antigens HBs), or C (antibody HCs), positive test for HIV, Treponema pallidum antibody positive.
5. Positive results from urine drug screen test.
6. Donate blood or lose blood 200 mL or more within 1 month prior to dosing.
7. Subjects who have used any medication, herbal medicine, nutritional supplements or health care products within 4 weeks prior to the first dose of study medication, or participated in other clinical studies or participated in a clinical study of test preparation within 3 months prior to the first dose of study medication.
8. History of needles or blood fainting, or have difficulty in blood collection, or cannot tolerate venipuncture for blood collection.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-08-02 (Estimated); Primary Completion 2023-01-04 (Estimated); Study Completion 2023-01-04 (Estimated)

PRIMARY OUTCOMES:
PK data for 14C-XZP-3287: Cmax | up to 15 days
  Maximum observed concentration for XZP-3287 in plasma and whole blood total radioactivity
PK data for 14C-XZP-3287: AUClast | up to 15 days
  Area under the plasma concentration time profile from time 0 to time of the last quantifiable concentration for XZP-3287 in plasma and whole blood total radioactivity
PK data for 14C-XZP-3287: AUCinf | up to 15 days
  Area under the plasma concentration time profile from time 0 to infinity for XZP-3287 in plasma and whole blood total radioactivity
PK data for 14C-XZP-3287: Tmax | up to 15 days
  Time of maximum observed concentration for XZP-3287 in plasma and whole blood total radioactivity
Quantitative analysis of cumulative excretion and excretion rate in excreta (urine and faeces) | up to 15 days
  Quantitative analysis of total radioactivity in excreta after oral [14C]XZP-3287 in healthy subjects, obtaining body material balance data and main excretion pathways

SECONDARY OUTCOMES:
Cmax of XZP-3287 in plasma | up to 15 days
  Maximum observed concentration for XZP-3287 in plasma
AUClast of XZP-3287 in plasma | up to 15 days
  Area under the plasma concentration time profile from time 0 to time of the last quantifiable concentration for XZP-3287 in plasma
AUCinf of XZP-3287 in plasma | up to 15 days
  Area under the plasma concentration time profile from time 0 to infinity for XZP-3287 in plasma
Tmax of XZP-3287 in plasma | up to 15 days
  Time of maximum observed concentration for XZP-3287 in plasma
To evaluate the safety of [14C] XZP-3287 | up to 29 days
  Percentage of Participants with Adverse Events (AEs)

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Gaobo Boren Hospital, Beijing, Beijing Municipality, China